CLINICAL TRIAL: NCT00380705
Title: Quality of Life in Asthma and Rhinitis Allergic With Singulair
Brief Title: Quality of Life in Asthma and Rhinitis Allergic With Singulair (0476-365)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0476-365; 2006_033
Record Dates: First submitted 2006-09-22; First posted 2006-09-26 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-01

CONDITIONS: Asthma; Rhinitis Allergic
MeSH Terms: conditions — Asthma; Rhinitis, Allergic, Perennial | interventions — montelukast; Duration of Therapy

INTERVENTIONS:
Drug: MK0476, Singulair, montelukast sodium / Duration of Treatment: 8 Weeks

SUMMARY:
Allow physicians not familiar with anti-leukotriene based therapy to test it

ELIGIBILITY:
Inclusion Criteria:

* Establish diagnosis of mild to moderate chronic asthma and/or allergic rhinitis currently on treatment
* Voluntary acceptance to participate in the study

Exclusion Criteria:

* Patients with cystic fibrosis
* Patients with known hypersensitivity to singulair or any of its components
* Patients with severe chronic asthma

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2005-03-18 (Actual); Primary Completion 2005-07-29 (Actual); Study Completion 2005-07-29 (Actual)

PRIMARY OUTCOMES:
Quality of life measures

SECONDARY OUTCOMES:
Nocturnal wake up, work or school absences, physical activity and recurrence of asthma and/or rhinitis

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC